CLINICAL TRIAL: NCT06596590
Title: Modified Water Vapor Thermal Therapy (REZUM) in Management of Patients With Large-volume Benign Prostatic Hyperplasia
Brief Title: Modified Water Vapor Thermal Therapy in Management of Patients With Large-volume Benign Prostatic Hyperplasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-SR-102
Record Dates: First submitted 2024-04-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Modified Water Vapor Thermal Therapy (REZUM) in Management of Patients With Large-volume Benign Prostatic Hyperplasia. The modified methods mainly include ablation optimization and combined imaging techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Modified Water Vapor Thermal Therapy (Experimental): The Rezum System is designed to treat patients with urinary symptoms associated with large volume BPH.
  Interventions: Device: Rezum

INTERVENTIONS:
Device: Rezum — The Rezum System is designed to treat patients with urinary symptoms associated with BPH. The Rezum System utilizes radiofrequency current to generate thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate in controlled 9-second doses. The vapor injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue, and the stored thermal energy is released, denaturing the cell membranes and causing cell death.

SUMMARY:
Water vapor thermal therapy (Rezum) is a minimally invasive treatment for benign prostatic hyperplasia (BPH) that uses injections of sterile water vapor directly into the prostate for tissue ablation. Although Rezum is currently indicated for use in men with prostate sizes ≥30 and ≤80 ml, the guidelines offer no recommendation with regards to Rezum therapy for those with large-volume glands.

DETAILED DESCRIPTION:
For prostates larger than 80ml, open or transurethral anatomical enucleation is recommended. Open prostatectomy has a higher risk of bleeding and slower postoperative recovery, with a higher probability of requiring blood transfusion. The incidence of urinary incontinence after transurethral enucleation ranges from 3.33% to 20%, possibly due to excessive traction and compression on the external urethral sphincter, leading to partial muscle fiber rupture. The rate of erectile dysfunction after enucleation is 8.82%, while retrograde ejaculation occurs in 6.37% of cases, especially for patients with larger prostates. Once these complications occur, they are often difficult to recover from and severely impact the patient's quality of life. In our center, the technique of Rezum has been further improved by incorporating ultrasound and MRI imaging guidance. The investigators design a reasonable and comprehensive ablation plan that ensures accurate positioning of enlarged prostate glands for complete and thorough ablation while ensuring efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 45 years of age who have obstructive symptoms secondary to BPH requiring invasive intervention.
2. IPSS score of ≥ 13.
3. Qmax: Peak flow rate ≤ 15 ml/sec.
4. Post-void residual (PVR) < 300 ml.
5. Prostate volume between 80 to 120 ml.
6. Subject able to complete the study protocol in the opinion of the Principal Investigator.

Exclusion Criteria:

1. History of any illness or surgery that in the opinion of the Principal Investigator may confound the results of the study.
2. Any prior minimally invasive intervention or surgical intervention for the symptoms of BPH.
3. Currently enrolled in another clinical trial.
4. Confirmed or suspected malignancy of prostate or bladder.
5. Documented active urinary tract infection by culture or bacterial prostatitis.
6. Neurogenic bladder or sphincter abnormalities.
7. Urethral strictures, bladder neck contracture or muscle spasms.
8. Bleeding disorder (note that use of anti-platelet medication is not an exclusion criterion).
9. Subjects who are interested in maintaining fertility.
10. Significant urge incontinence.
11. Unable or unwilling to sign the Informed Consent Form.
12. Any cognitive disorder that interferes with or precludes a subject from directly and accurately communicating with the Principal Investigator regarding the study.

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) change from baseline to 3 months. | from baseline to 3 months
  International prostate symptom score (IPSS) is a questionnaire used to indicate the severity of LUTS symptoms, There are 7 questions relating to different symptoms subjects be experiencing. 7 questions about patients' urinating include Incomplete emptying, Frequency, Intermittency, Urgency, Weak stream, Straining and Nocturia, every question have 0-5 scores according to Prostate Symptom, the higher score mean patient have more severe the symptoms.
  IPSS total score: the minimum score is 0 and maximum score are 35. IPSS total 0-7 scores are mild symptoms, IPSS total 8-19 scores are moderate symptoms and IPSS total 20-35 scores are severe symptoms. International Prostate Symptom Score (IPSS) scores were recorded at baseline to 3 months. The mean change in IPSS was calculated.

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) change from baseline to 1 month, 3 months, 6 months, 1 year, then annually to 3 years. | 1 month, 3 months, 6 months, 1 year, then annually to 3 years
  International prostate symptom score (IPSS) is a questionnaire used to indicate the severity of LUTS symptoms, There are 7 questions relating to different symptoms subjects be experiencing. 7 questions about patients' urinating include Incomplete emptying, Frequency, Intermittency, Urgency, Weak stream, Straining and Nocturia, every question have 0-5 scores according to Prostate Symptom, the higher score mean patient have more severe the symptoms.
  IPSS total score: the minimum score is 0 and maximum score are 35. IPSS total 0-7 scores are mild symptoms, IPSS total 8-19 scores are moderate symptoms and IPSS total 20-35 scores are severe symptoms. International Prostate Symptom Score (IPSS) scores were recorded at baseline to 1 month, 3 months, 6 months, 1 year, then annually to 3 years. The mean change in IPSS was calculated.
The change of peak flow rate (Qmax) | 1 month, 3 months, 6 months, 1 year, then annually to 3 years
Post void residual urine volume (PVR） | 1 month, 3 months, 6 months, 1 year, then annually to 3 years
Quality of life (QoL) | 1 month, 3 months, 6 months, 1 year, then annually to 3 years
  There is only 1 question about Quality of life due to urinary symptoms which is 'If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?' This question have 0-6 scores according to patient's satisfaction about Quality of Life, the higher score mean patient have poor satisfaction.
  The change was the baseline value minus the value at 1 month, 3 months, 6 months, 1 year, then annually to 3 years.
Ejective function (MSHQ-EjD) | 1 month, 3 months, 6 months, 1 year, then annually to 3 years
  Ejective function (MSHQ-EjD) is a questionnaire used to assess the ejective function. There are 4 questions relating to Ejaculation dysfunction which need patients to answer. 3 questions about patients' ejective function assessing include completion of ejaculation, Strength of ejaculation and Volume of semen when ejaculation. Every question have 0-5 scores according to assessing the ejective function, the lower score mean patient have more severe the ejective function.
  MSHQ-EjD total score: the minimum score is 0 and maximum score are 15. The change are the value at 1 month, 3 months, 6 months, 1 year, then annually to 3 years minus value at baseline.
The change of International Index of Erectile Function (IIEF) | 1 month, 3 months, 6 months, 1 year, then annually to 3 years
  Erectile Function(IIEF) is a questionnaire used to assess the Sexual Health Inventory of men. There are 5 questions relating to Erectile Function which need patients to answer. Every question have 0-5 scores, the lower score mean patient have more severe the Erectile Function.
  The IIEF-5 is administered as a screening instrument for the presence & severity of ED in conjunction with the clinical assessment. The score is the sun of the responses to the five items, so that overall score may range from 0 to 25. A score of 20 or higher indicates a normal degree of erectile functioning. Low scores (10 or less) indicate moderate to severe ED.
  The change are the value at 1 month, 3 months, 6 months, 1 year, then annually to 3 years minus value at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, PhD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China